CLINICAL TRIAL: NCT07312383
Title: Skin Microcirculation in Patients With Lower Limb Atherosclerosis
Acronym: SMILLA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ODI Medical AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIV-NO-25-10-054857
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Percutaneous Transluminal Angioplasty; Atherosclerosis of Arteries of the Extremities, Unspecified
Keywords: Atherosclerosis; Lower leg ischaemia; PTA
MeSH Terms: conditions — Atherosclerosis | interventions — Physical Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients scheduled for elective PTA (Other)
  Interventions: Device: Examination with the ODI-Tech medical device

INTERVENTIONS:
Device: Examination with the ODI-Tech medical device — Diffuse reflectance spectroscopy and computer-assisted microscopy.

SUMMARY:
The aim of this study is to explore the ability of the non-invasive device ODI-Tech® to monitor changes in microvascular blood flow in patients with lower limb ischemia undergoing the procedure percutaneous transluminal angioplasty (PTA). Microvascular data from patients and healthy case matched controls at baseline will be compared.15 patients and 15 healthy case matched controls will be enrolled.

DETAILED DESCRIPTION:
This clinical investigation is designed as a prospective study of limb skin nutritive capillary perfusion and oxygen extraction in patients with lower limb atherosclerosis and severe symptoms before and following elective PTA.

15 patients with critical lower limb atherosclerosis and ischemia in Rutherford grade 3 - 6 undergoing PTA, as well as 15 healthy case matched controls will be enrolled. Measurements will be performed at baseline, prior to PTA, immediately after PTA, 1 day and 30 days post PTA. Healthy case matched controls will be measured at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Lower limb atherosclerosis and ischemia in Rutherford grade 3-6
* Obstructive infra-inguinal arterial lesions combined with open distal part of the anterior tibial artery
* Scheduled for elective PTA
* Able to give informed consent

Exclusion Criteria:

* Active skin infection at the region of interest (site to be examined, dorsum of hand and foot)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Changes in skin microvascular oxygen saturation (SmvO2) | From baseline to 40 days post PTA
Changes in functional Capillary Density (FCD) | From baseline to 40 days post PTA.

SECONDARY OUTCOMES:
Incidence of AE/ADE/SAE/SADE/DD | From baseline to 40 days post PTA

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data supporting the results of the study.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: From 6 months after publication of the primary results and until 5 years thereafter.
Access Criteria: De-identified data will be made available to qualified researchers who submit a scientific and methodologically sound proposal to the sponsor.

REFERENCES:
- [Background] Mork C, Kvernebo K, Asker CL, Salerud EG. Reduced skin capillary density during attacks of erythromelalgia implies arteriovenous shunting as pathogenetic mechanism. J Invest Dermatol. 2002 Oct;119(4):949-53. doi: 10.1046/j.1523-1747.2002.00218.x. PMID 12406343
- [Background] Wester T, Awan ZA, Kvernebo TS, Salerud G, Kvernebo K. Skin microvascular morphology and hemodynamics during treatment with veno-arterial extra-corporeal membrane oxygenation. Clin Hemorheol Microcirc. 2014;56(2):119-31. doi: 10.3233/CH-131670. PMID 23357861
- [Background] Fredly S, Fugelseth D, Nygaard CS, Salerud EG, Stiris T, Kvernebo K. Noninvasive assessments of oxygen delivery from the microcirculation to skin in hypothermia-treated asphyxiated newborn infants. Pediatr Res. 2016 Jun;79(6):902-6. doi: 10.1038/pr.2016.16. Epub 2016 Feb 8. PMID 26854800
- [Background] Sundheim LK, Sporastoyl AH, Wester T, Salerud G, Kvernebo K. Acute skin trauma induces hyperemia, but superficial papillary nutritive perfusion remains unchanged. Microcirculation. 2017 Oct;24(7). doi: 10.1111/micc.12389. PMID 28632939